CLINICAL TRIAL: NCT02757001
Title: Inferior Vena Cava Retrievable Filters: Spanish Register (REFiVeC)
Brief Title: Inferior Vena Cava Retrievable Filters: Spanish Register
Acronym: REFiVeC
Status: Completed | Type: Observational
Sponsor: Group of Research in Minimally Invasive Techniques (Other)
Collaborators: SERVEI (Sociedad Española de Radiología Vascular e Intervencionista) (Unknown)
Responsible Party: Sponsor
Other Study IDs: GITMI
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2019-07

CONDITIONS: Vena Cava Filters
Keywords: Retrievable Inferior Vena Cava Filters; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Inferior vena cava filter placement and retrieval — There are really no interventions in this study. This is an prospective observational study of patients that have been implanted a inferior vena cava filter with intention to be retrieved.
  Patients are recruited when the filter is implanted, and the investigators observe when is it finally retrieved, and if there is any complication at the retrieval of the filter.

SUMMARY:
Spanish registry of retrievable vena cava filters.

This registry is sponsored by the Spanish Society of Vascular and Interventional Radiology (SERVEI) and conducted by the Research Group GITMI (Group of Research in Minimally Invasive Techniques) of the University of Zaragoza (Spain).

A software tool hosted on the official website of SERVEI and the journal Intervencionismo will be used for data collection a(https://estudios.watsoncme.com).

DETAILED DESCRIPTION:
This is an prospective observational study of patients that have been implanted a inferior vena cava filter with intention to be retrieved.

Patients are recruited when the filter is implanted, and the investigators observe when is it finally retrieved (dwell time), if retrieval is possible or not, and if there is any complication at the retrieval of the filter.

ELIGIBILITY:
Inclusion Criteria:

* Indicated inferior vena cava filter implantation
* Signed informed consent

Exclusion Criteria:

* Permanent filters (including retrievable filters intended to be used as permanent ones)
* Impossibility of follow-up (3, 6 and 12 months)
* Life expectancy less than a year
* Patient refusal to be included in the study, at any time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom a vena cava filter has been implanted with intention of being retrieved (non-permanent).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Success of retrieval | 12 months
  The primary outcome of this study is to verify if the filter can be retrieved on the scheduled day of retrieval (yes/no).

SECONDARY OUTCOMES:
Dwell time | 12 months
  Final dwell time of the filter (number of days from implantation to retrieval). It will be compared to the expected dwell time at the time of implantation.
Complications in retrieval | 12 months
  Difficulties in retrieval and complications at the time of retrieval will be specifically recorded.
Overall adverse events | 12 months
  Registry of adverse events from filter implantation until retrieval.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A De Gregorio, Ph.D., Principal Investigator — Minimal Invasive Techniques Research Group
Locations (6):
- Spain (6):
  - Hospital de Basurto, Bilbao
  - Hospital Universitario La Princesa, Madrid
  - Hospital Vithas Nisa Pardo de Aravaca, Madrid
  - Hospital Regional Carlos Haya, Málaga
  - Hospital Universitario Rio Hortega, Valladolid
  - Lozano Blesa University Hospital, Zaragoza